CLINICAL TRIAL: NCT05720741
Title: Project THINK: Testing a Single-Session, Digital Cognitive Restructuring Intervention for Youth Mental Health in a Randomized Controlled Trial
Brief Title: Project THINK: Trial of a Brief Cognitive Restructuring Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Joshua Steinberg, Principal Investigator, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB22-1364
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Anxiety; Depression; Stress
Keywords: digital; mental health intervention
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Participants (anticipated N=1,625), ages 10-16 years, will be randomized to complete one 30-minute, digital programs: (1) Project THINK: a program designed to teach adolescents how to identify and modify unhelpful thoughts; or (2) Project SHARE: a control program designed to teach adolescents to identify and share emotions with trusted adults. A priori power analyses revealed that N=788 participants are needed to detect a small effect size (.2, the approximate effect size found in recent brief digital intervention RCTs) using two-tailed tests with α = .05. In line with findings from similar studies, attrition in online survey studies with students is high; a recent meta-analysis of ~1,000 studies that used online assessments found a mean attrition rate of 51.5%. Assuming this level of attrition, to achieve the desired sample (N=788), the most conservative estimate of the minimum number of participants needed is 1,625 students at baseline.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project THINK (Experimental): Project THINK is a 30-minute self-guided digital intervention designed to teach children and adolescents how to change the way that they think. Specifically, Project THINK is based on the principles of cognitive restructuring, a core component of cognitive behavioral therapy, a gold standard treatment for internalizing disorders. Project THINK uses vignettes, interactive activities, and engaging graphics to teach youth a systematic strategy for assessing the presence of unhelpful thoughts and replacing them with more helpful ones. Although not yet formally tested in a randomized trial, Project Think has been used by hundreds of students, and feedback has been very positive.
  Interventions: Behavioral: Project THINK
- Project SHARE (Placebo Comparator): Intervention delivered in a web browser that focuses on encouraging feelings disclosure to trusted others using facts about the brain, testimonials from peers, and writing exercises (also referred to as Sharing Feelings Intervention; Schleider et al., 2021).
  Interventions: Behavioral: Project SHARE

INTERVENTIONS:
Behavioral: Project THINK — Project THINK is a 30-minute self-guided digital intervention designed to teach children and adolescents how to change the way that they think. Specifically, Project THINK is based on the principles of cognitive restructuring, a core component of cognitive behavioral therapy, a gold standard treatment for internalizing disorders. Project THINK uses vignettes, interactive activities, and engaging graphics to teach youth a systematic strategy for assessing the presence of unhelpful thoughts and replacing them with more helpful ones. Although never formally tested in a randomized trial, Project Think has been used by hundreds of students, and feedback has been very positive.
  Arms: Project THINK
Behavioral: Project SHARE — Intervention delivered in a web browser that focuses on encouraging feelings disclosure to trusted others using facts about the brain, testimonials from peers, and writing exercises (also referred to as Sharing Feelings Intervention; Schleider et al., 2021).
  Arms: Project SHARE

SUMMARY:
This project will involve testing a brief (~30 minute) digital intervention aimed at teaching youth the evidence-based strategy of changing unhelpful thoughts (i.e., cognitive restructuring). The investigators will test the intervention's efficacy compared to an active control condition. Participants (students in grades 5-10 in U.S. schools) will be asked to complete measures of mental health and well-being prior to the intervention as well as 1, 3, and 6-months after the intervention. If the intervention is found to be effective, its brevity and scalability would make it an invaluable resource for supplementing traditional psychotherapy and potentially preventing the onset of mental illness requiring specialized intensive care.

DETAILED DESCRIPTION:
More than one in five adolescents will experience at least one mental health disorder requiring treatment; however, 75% of these adolescents will never receive mental health care, in large part due to the fact that there are far fewer trained clinicians than are necessary to address growing youth mental healthcare needs. Furthermore, the disparity between the number of available clinicians and those in need of mental health services is increasing. Between 2016 and 2020, the number of American children ages 3-17 diagnosed with an anxiety disorder or depression grew by 29% and 27%, respectively, whereas the American Psychological Association (APA) reports that the number of clinicians treating youth has continued to remain low, with only 4,000 out of 100,000 U.S. clinical psychologists identifying as child and adolescent clinicians. One possible solution to this issue of treatment access is to emphasize prevention and intervention strategies that can help reduce the number of young people who may develop mental health problems requiring more intensive care. However, even such prevention efforts have historically required large amounts of human capital for implementation. Fortunately, in recent years, digital mental health interventions have emerged as a potential solution to this issue as they offer scalable and cost-effective ways of preventing and intervening on mental health problems. Digital interventions requiring little-to-no professional support are especially appealing because they are easy to implement. Further, digital mental health interventions have been found to be efficacious for common mental health problems such as depression and anxiety, and some are effective for young people even in a single session.

The investigators propose one such intervention utilizing technology to address issues of access to mental health resources: Project THINK is a 30-minute self-guided digital intervention designed to teach children and adolescents how to change the way that they think. Specifically, Project THINK is based on the principles of cognitive restructuring, a core component of cognitive behavioral therapy, a gold standard treatment for internalizing disorders. Project THINK uses vignettes, interactive activities, and engaging graphics to teach youth a systematic strategy for assessing the presence of unhelpful thoughts and replacing them with more helpful ones. Although not yet formally tested in a randomized trial, Project Think has been used by hundreds of students, and feedback has been very positive.

Aim 1. In collaboration with U.S. middle schools, the investigators aim to conduct a randomized trial examining the efficacy of Project THINK relative to an active control condition, Project SHARE (i.e., Sharing Feelings)-which teaches users to identify their emotions and share them with trusted adults-on improving symptoms of mental health and well-being among adolescents. The investigators aim to recruit 1,625 participants in grades 5-10 (ages 10-16 years). According to a priori power analyses and after accounting for high expected attrition, this target sample size will provide sufficient power (1-β; 80%) to detect overall mean group differences and moderation effects of small effect size (.2; minimum N=788) using two-tailed tests with α = .05. The use of Project SHARE is appropriate in this context given that it has been used in past research studies and it has been found to be useful for young people, but it is not designed to target symptoms of psychopathology.

During a time selected by school partners (likely to be a wellness/physical education/gym class), participating students will choose whether they will assent to participate in the study. Only those participants whose parents have not elected to opt their child out of the study beforehand will be asked if they would like to participate. If students assent via an online form, they will be directed to an online battery of validated measures focused on mental health and well-being (e.g., Behaviors and Feelings Survey, and the Emotion Regulation Questionnaire--Child/Adolescent Version-Cognitive Reappraisal Subscale). Students will then be randomized to complete the Project THINK intervention or the Project SHARE active control online program; these two programs are similar in length and format. Immediately following completion of one of the two programs, participants will be asked to answer online demographic questions and to provide feedback on the intervention's helpfulness. All study procedures will be conducted via Qualtrics, and the investigators will conduct separate analyses for the subsample of students with elevated symptoms of psychopathology at baseline to assess the potentially different effects of Project THINK as a universal versus indicated prevention program.

Aim 2. The investigators aim to examine the effects of Project THINK relative to Project SHARE over time. Toward this end, participating students will be asked to complete a battery of measures at three follow-up timepoints: 1-month, 3-months, and 6-months after the baseline assessment and intervention administration. These follow-up measures represent a subset of the measures assessed at baseline (i.e., all measures assessed at baseline except demographic questions and feedback regarding intervention helpfulness). Once more, the investigators will conduct separate analyses for the subsample of students with elevated symptoms of psychopathology at the baseline assessment.

A secondary aim of this study is to interview a subset of student participants (10-30) from one of the partner schools. Following the one-month follow-up survey, the investigators will select an equal number of participants who are either 'responders' or 'not responders' to the Project THINK intervention. 'Responders' will be operationalized as those who were randomized to Project THINK and experienced a decline in internalizing symptoms (as measured by the Behavior and Feelings Survey). 'Non-responders' will be operationalized as those whose internalizing symptoms are not reduced. Through a semi-structured interview and thematic analysis in NVivo software, the investigators aim to identify patterns or themes that emerge in participants' experiences, and then examine whether these themes differ based on differential symptom trajectories. The investigators aim to examine the participants' recall of intervention content, comprehension of skills, perceived relevance of the skills, ways they used the skills following the intervention, as well as overall thoughts on the intervention and its delivery (sample questions are below). The participants who are selected for the interview will be excluded from the primary analyses at the 3 and 6-month follow-ups due to the potential interventional effects of the interview.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescent is in grades 5-10 (inclusive) at partnering schools
2. Adolescent is between the ages of 10 through 16 years (inclusive) at the time of study enrollment
3. Adolescent and at least one guardian consent to adolescent participation in study
4. Adolescent reads English well enough to effectively complete the digital programs
5. Adolescent has access to a digital device

Exclusion Criteria:

1. Adolescent is non-English speaking, as the programs are only available in English
2. Adolescent does not have access to a digital device
3. Adolescent has an intellectual disability that precludes comprehension of the program content

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 597 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Behavior and Feelings Survey (Internalizing Subscale) from Baseline to 1-month Follow-up | Baseline to 1-month follow-up
  Trajectories of self-reported symptoms of anxiety and depression from the 6-item (each item rated on a 0-4 scale, with higher ratings indicating more symptoms) Internalizing subscale of the Behavior and Feelings Survey. Total scores range from 0 to 24, with higher scores indicating more symptoms.
Change in Behavior and Feelings Survey (Internalizing Subscale) from Baseline to 3-month Follow-up | Baseline to 3-month follow-up
  Trajectories of self-reported symptoms of anxiety and depression from the 6-item (each item rated on a 0-4 scale, with higher ratings indicating more symptoms) Internalizing subscale of the Behavior and Feelings Survey. Total scores range from 0 to 24, with higher scores indicating more symptoms.
Change in Behavior and Feelings Survey (Internalizing Subscale) from Baseline to 6-month Follow-up | Baseline to 6-month follow-up
  Trajectories of self-reported symptoms of anxiety and depression from the 6-item (each item rated on a 0-4 scale, with higher ratings indicating more symptoms) Internalizing subscale of the Behavior and Feelings Survey. Total scores range from 0 to 24, with higher scores indicating more symptoms.

SECONDARY OUTCOMES:
Perceived Program Acceptability and Helpfulness | Immediately post-intervention
  Post-intervention feedback on the program's perceived acceptability and helpfulness as measured via a 7-item scale, with each item rated on a 1-5 scale, with higher scores indicating greater acceptability and helpfulness.
Change in Behavior and Feelings Survey (Externalizing Subscale) from Baseline to 1-month Follow-up | Baseline to 1-month follow-up
  Trajectories of self-reported misbehavior from the 6-item (each item rated on a 0-4 scale, with higher ratings indicating more symptoms) Externalizing subscale of the Behavior and Feelings Survey. Total scores range from 0 to 24, with higher scores indicating more symptoms.
Change in Behavior and Feelings Survey (Externalizing Subscale) from Baseline to 3-month Follow-up | Baseline to 3-month follow-up
  Trajectories of self-reported misbehavior from the 6-item (each item rated on a 0-4 scale, with higher ratings indicating more symptoms) Externalizing subscale of the Behavior and Feelings Survey. Total scores range from 0 to 24, with higher scores indicating more symptoms.
Change in Behavior and Feelings Survey (Externalizing Subscale) from Baseline to 6-month Follow-up | Baseline to 6-month follow-up
  Trajectories of self-reported misbehavior from the 6-item (each item rated on a 0-4 scale, with higher ratings indicating more symptoms) Externalizing subscale of the Behavior and Feelings Survey. Total scores range from 0 to 24, with higher scores indicating more symptoms.
Change in Emotion Regulation Questionnaire--Child/Adolescent Version (Cognitive Reappraisal Subscale) from Baseline to 1-month follow-up | Baseline to 1-month follow-up
  Trajectories of self-reported tendency to regulate emotions using cognitive reappraisal strategies from the 6-item (each item rated on a 1 to 7 scale with 7 indicating more use of cognitive reappraisal emotion regulation strategies) Cognitive Reappraisal Facet of the Emotion Regulation Questionnaire.
Change in Emotion Regulation Questionnaire-Child/Adolescent Version (Cognitive Reappraisal Subscale) from Baseline to 3-month follow-up | Baseline to 3-month follow-up
  Trajectories of self-reported tendency to regulate emotions using cognitive reappraisal strategies from the 6-item (each item rated on a 1 to 7 scale with 7 indicating more use of cognitive reappraisal emotion regulation strategies) Cognitive Reappraisal Facet of the Emotion Regulation Questionnaire.
Change in Emotion Regulation Questionnaire--Child/Adolescent Version (Cognitive Reappraisal Subscale) from Baseline to 6-month follow-up | Baseline to 6-month follow-up
  Trajectories of self-reported tendency to regulate emotions using cognitive reappraisal strategies from the 6-item (each item rated on a 1 to 7 scale with 7 indicating more use of cognitive reappraisal emotion regulation strategies) Cognitive Reappraisal Facet of the Emotion Regulation Questionnaire.
Treatment Expectancy Measure | Immediately pre-intervention
  Treatment expectations will be assessed at pre-intervention via a novel 4-item measure (0-10 scale) evaluating participants' expectations of intervention effects.

OTHER OUTCOMES:
Qualitative Responses via Semi-Structured Interview | Between the 1 and 3-month follow-ups
  Questions including but not limited to the following:
  * What can you recall about the contents of the Project THINK intervention?
  * How have you used the skills taught in the Project THINK intervention? If so, how have you used them? Can you give me some examples of times you used it or felt like you could use it (what stopped you from using the skills learned)?
  * How relevant is the content of Project THINK to your life?
  * What was your understanding of what Project Think was trying to teach?
  * What did you find helpful about Project THINK?
  * What did you find unhelpful about Project THINK?
  * Did you like doing the intervention online?
  * Did you like this format of delivery? Or are there other ways you wish you could access this?
  * Did you have any expectations of what the intervention might do? If so, were they met?
  * How did you feel doing the intervention? Was it a positive/negative experience for you?
  * What are some ways we could change for you to use it more?

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Analytic code will be made available upon publication of trial results. Study protocol and SAP are available with this registration submission.

REFERENCES:
- See also: Statistical Analysis Plan — https://docs.google.com/document/d/1yGx6BODExiSHRqO0EG-MSIX6Qf4QB2BNZUIB14QrKCQ/edit?usp=sharing